CLINICAL TRIAL: NCT03779178
Title: Microcirculatory and Macrocirculatory Effects of Landiolol in Prevention of Postoperative Atrial Fibrillation: a Randomized Study.
Brief Title: Landiolol in Postoperative Atrial Fibrillation
Acronym: MMELPOAF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL16_0743; 2018-000307-17 (EudraCT Number)
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: landiolol; microcirculation; cardiac surgery; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — landiolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landiolol group (Experimental): Landiolol perfusion in incremental doses (range 0.5 to 10 µg/kg/min) over 2 hours
  Interventions: Drug: Landiolol
- Placebo group (Placebo Comparator): Placebo perfusion in incremental doses (range 0.03 to 0.6 mL/kg/h) over 2 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Landiolol — Landiolol perfusion over 120 minutes in incremental doses : 0.5, 1, 2, 5 and 10 µg/kg/min. Doses are modified every 20 minutes
  Arms: Landiolol group
Drug: Placebo — Placebo perfusion is sodium chloride NaCl 0.9% over 120 minutes in incremental doses : 0.03, 0.06, 0.12, 0.3 and 0.6 mL/kg/h. Doses are modified every 20 minutes. Perfusion are similar in landiolol group to preserve blind.
  Arms: Placebo group

SUMMARY:
Postoperative atrial fibrillation is a common complication after cardiac surgery and is associated with an elevation of morbidity and mortality. The recommended treatment includes heart rate control with a beta blocker. Landiolol is a new-generation beta-blocker with favourable pharmacologic properties making an interesting drug to treat postoperative atrial fibrillation. However, Landiolol micro and macrocirculatory effects in the setting of atrial fibrillation are yet to describe. The aim of this study is to describe microcirculatory effects of incremental doses of landiolol in postoperative atrial fibrillation compared to a placebo. Our hypothesis is Landiolol will improve microcirculation disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent conventional cardiac surgery
* Age > 18 years
* Writing contentment

Exclusion Criteria:

* Pre-existing chronic atrial fibrillation
* Contraindication to beta-blockers
* Circulatory shock (cardiac index<2.2 L/min and lactate>4mmol/L)
* Distributive shock (cardiac index>2.2 L/min with norepinephrine dose > 0.3 µg/kg/min to reach mean arterial pressure > 65mmHg).
* Acute respiratory distress
* Major bleeding (>200mL/h)
* Patient already included into an interventional clinical study
* Pregnancy
* No social security insurance
* Patient not able to give consent (curators, patients deprived of public rights)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Tissular resaturation speed measured by somatic near-infrared spectroscopy (NIRS) | at 20 minutes
  Tissular resaturation speed is measured after vascular occlusion test. At each time end-point, an occlusion of the arm blood flow with a tourniquet is made. After the nadir of the tissular saturation of the arm is reached the tourniquet is released and the resaturation speed is measured using the NIRS.
Tissular resaturation speed measured by somatic near-infrared spectroscopy (NIRS) | at 40 minutes
  Tissular resaturation speed is measured after vascular occlusion test. At each time end-point, an occlusion of the arm blood flow with a tourniquet is made. After the nadir of the tissular saturation of the arm is reached the tourniquet is released and the resaturation speed is measured using the NIRS.
Tissular resaturation speed measured by somatic near-infrared spectroscopy (NIRS) | at 60 minutes
  Tissular resaturation speed is measured after vascular occlusion test. At each time end-point, an occlusion of the arm blood flow with a tourniquet is made. After the nadir of the tissular saturation of the arm is reached the tourniquet is released and the resaturation speed is measured using the NIRS.
Tissular resaturation speed measured by somatic near-infrared spectroscopy (NIRS) | at 80 minutes
  Tissular resaturation speed is measured after vascular occlusion test. At each time end-point, an occlusion of the arm blood flow with a tourniquet is made. After the nadir of the tissular saturation of the arm is reached the tourniquet is released and the resaturation speed is measured using the NIRS.
Tissular resaturation speed measured by somatic near-infrared spectroscopy (NIRS) | at 100 minutes
  Tissular resaturation speed is measured after vascular occlusion test. At each time end-point, an occlusion of the arm blood flow with a tourniquet is made. After the nadir of the tissular saturation of the arm is reached the tourniquet is released and the resaturation speed is measured using the NIRS.
Tissular resaturation speed measured by somatic near-infrared spectroscopy (NIRS) | at 120 minutes
  Tissular resaturation speed is measured after vascular occlusion test. At each time end-point, an occlusion of the arm blood flow with a tourniquet is made. After the nadir of the tissular saturation of the arm is reached the tourniquet is released and the resaturation speed is measured using the NIRS.

SECONDARY OUTCOMES:
Microcirculatory mean flow index (MIF) acquired by sublingual microscopy | at 120 minutes
proportion of perfused vessels acquired by sublingual microscopy | at 120 minutes
functional capillary density acquired by sublingual microscopy | at 120 minutes
De Backer score acquired by sublingual microscopy | at 120 minutes
heterogeneity of the mean flow index acquired by sublingual microscopy | at 120 minutes
Heart rate | at 120 minutes
  hemodynamic parameters
systolic arterial pressure | at 120 minutes
  hemodynamic parameters
diastolic arterial pressure | at 120 minutes
  hemodynamic parameters
cardiac output measured by transthoracic echocardiography | at 120 minutes
  hemodynamic parameters
systemic vascular resistance | at 120 minutes
  hemodynamic parameters
arterial elastance. | at 120 minutes
  hemodynamic parameters
Ejection fraction of the left ventricle (FEVG) | at 120 minutes
  echocardiographic parameters
telesystolic volumes of the right ventricle | at 120 minutes
  echocardiographic parameters
telesystolic volumes of the left ventricle | at 120 minutes
  echocardiographic parameters
telediastolic volumes of the right ventricle | at 120 minutes
  echocardiographic parameters
telediastolic volumes of the left ventricle | at 120 minutes
  echocardiographic parameters
right ventricle contractility (measured with TAPSE and tricuspid S-wave) | at 120 minutes
  echocardiographic parameters
intracardiac filling pressure profiles (E/a, E/Vp, E/e') | at 120 minutes
  echocardiographic parameters
oxygen consumption (V02) | at 120 minutes
  tissular perfusion parameters
oxygen delivery (DO2), | at 120 minutes
  tissular perfusion parameters
carbon dioxide production (VCO2) | at 120 minutes
  tissular perfusion parameters
arterial lactate | at 120 minutes
  tissular perfusion parameters

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Jacquet-Lagrèze, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel, Bron, France

REFERENCES:
- [Result] Ferraris A, Jacquet-Lagreze M, Cazenave L, Fornier W, Jalalzai W, Rousseau-Saine N, Allaouchiche B, Junot S, Pozzi M, Fellahi JL; Anesthesie-Reanimation Coeur-Thorax-Vaisseaux (ARCOTHOVA) Group. Microcirculatory effects of landiolol: a double-blind, randomised, controlled study after cardiac surgery. Br J Anaesth. 2021 Jun;126(6):e212-e214. doi: 10.1016/j.bja.2021.03.013. Epub 2021 Apr 24. No abstract available. PMID 33902917